CLINICAL TRIAL: NCT02399618
Title: Freeze-dried, Capsulized Fecal Microbiota Transplantation for Relapsing Clostridium Difficile Infection
Brief Title: Freeze-dried, Capsulized FMT for RCDI
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Ding Chao, MD candidate, Jinling Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Freeze-dried FMT-2015
Record Dates: First submitted 2015-03-21; First posted 2015-03-26 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Clostridium Difficile Infection
Keywords: Clostridium difficile Infection; Fecal Microbiota Transplantation; Freeze-dried; Acid-resistant Capsules
MeSH Terms: conditions — Clostridium Infections | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Capsulized freeze-dried FMT (Experimental): Reconstitution of normal flora with capsulized freeze-dried fecal inoculum
  Interventions: Drug: Fecal Microbiota Transplantation

INTERVENTIONS:
Drug: Fecal Microbiota Transplantation — Fecal microbiota transplant from healthy, unrelated donor via freeze-dried capsule
  Other Names: Fecal bacteriotherapy

SUMMARY:
Recurrent or refractory Clostridium difficile Infection (RCDI), with a recent increased incidence, is one of the most difficult and increasingly challenges for CDI. Since Fecal Microbiota Transplantation (FMT) has been accepted as the first-line therapy for RCDI, it is prudent to consider less invasive and more convenient means of administering FMT. The majority of reported FMT procedures have been performed with fresh or frozen stool suspensions via colonoscopy or nasojejunal tube. Nowadays, using acid-resistant hypromellose capsules, Youngster et al. significantly simplified the clinical practice of FMT and removed the need for invasive gastrointestinal procedures. However, to avoid undesirable disintegration, those capsules containing stool suspensions must be kept frozen all the time, which extremely limits their widespread application. The purpose of this study is to evaluate the efficacy and safety of freeze-dried, capsulized FMT for RCDI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractory, recurrent or relapsing C. difficile infection (RCDI), as defined in guidelines as a relapse of CDI after having at least 3 episodes of mild to moderate CDI and failure of a 6- to 8-week taper with vancomycin with or without an alternative antibiotic or at least 2 episodes of severe CDI resulting in hospitalization and associated with significant morbidity;
* Willingness to accept risk of healthy unrelated donor stool.

Exclusion Criteria:

* Delayed gastric emptying syndrome;
* Known chronic aspiration;
* Swallowing dysfunction or oral-motor dyscoordination;
* Pregnant or breast-feeding women;
* Usage of probiotics, prebiotics or synbiotics within the last month;
* Smoking or alcohol use within the last month;
* Patients with an exacerbation of condition not because of CDI;
* Patients on major immunosuppressive agents or with any other cause of severe immunodeficiency;
* Patients with a history of significant allergy because of diet;
* Patients on any agents affecting fecal bacteriology because of comorbidities.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Safety is assessed by clinical symptoms, exam, signs (GI and systemic). | Up to 3 months post-FMT
  Safety is assessed by clinical symptoms, exam, signs (GI and systemic).
Efficacy | Up to 3 months post-FMT
  Efficacy is defined as resolution of C. Difficile signs and symptoms off antibiotics for C. difficile.

SECONDARY OUTCOMES:
Change of fecal bacteriology | Up to 1 month post-FMT
  Fecal microbiology is characterized by 16S rRNA gene-based analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, MD, Study Director — Department of Generay Surgery, Jinling hosptal, Medical School of Nanjing University
Locations (1):
- Department of Generay Surgery, Jinling hosptal, Medical School of Nanjing University, Nanjing, Jiangsu, China